CLINICAL TRIAL: NCT03582085
Title: Phase II Clinical Trial: Multi-dosing the BCG Vaccine for Fibromyalgia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding at the current time.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Denise Louise Faustman, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18114
Record Dates: First submitted 2018-06-18; First posted 2018-07-10 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — BCG Vaccine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Half of the subjects will be placed in the multi-dose BCG group and half will be placed in the placebo group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bacillus Calmette-Guerin (BCG) (Experimental): 3 BCG vaccinations spaced 1 year apart.
  Interventions: Biological: Bacillus Calmette Guerin Vaccine
- Placebo Comparator: Saline injections (Placebo Comparator): 3 saline injections spaced 1 year apart.
  Interventions: Biological: Saline Injection

INTERVENTIONS:
Biological: Bacillus Calmette Guerin Vaccine — Experimental
  Other Names: BCG
  Arms: Bacillus Calmette-Guerin (BCG)
Biological: Saline Injection — Placebo
  Arms: Placebo Comparator: Saline injections

SUMMARY:
The investigators are doing this research study to explore whether the bacillus Calmette-Guérin (BCG) vaccine can be an effective treatment for fibromyalgia. The researchers believe that the BCG vaccine can benefit people with fibromyalgia by increasing immune signaling molecules, called cytokines. The Faustman Immunobiology Laboratory has previously studied BCG in long term type 1 diabetics, and found that BCG vaccinations showed a short and small pancreas effect of restored insulin secretion.

Eligible volunteers will be vaccinated with BCG in repeat fashion over a period of three years or receive placebo treatment. The investigators hypothesize that these repeat injections of BCG will reduce symptom severity by increasing immune signaling cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia
* HIV antibody negative
* Normal complete blood count (CBC), LFT, metabolic panel
* Meets the requirements for pain measured by the widespread pain index and symptom severity scale
* Negative pregnancy test within 7 days before initiation of study drug (Female only)

Exclusion Criteria:

* History of HIV or hepatitis
* History of tuberculosis, mycobacterium exposure, TB risk factors, positive interferon-gamma release assay (IGRA, also known as T-SPOT.TB test) or BCG vaccination
* Current treatment with glucocorticoids or disease likely to require steroid therapy
* Conditions or treatments associated with risk of infections such as patients with a previous history of severe burns, or treatment with immunosuppressive medications of any type
* Daily use of aspirin > 160 mg, or chronic, daily NSAIDs
* Current treatment with antibiotics
* History of keloid formation
* Severe pain due to other conditions
* Current treatment with any Type II diabetes medication (such as metformin, farxiga, etc.)
* Pregnant or not using acceptable birth control
* Living with someone who is immunosuppressed and/or at high risk for infectious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in overall fibromyalgia symptoms since beginning the clinical trial, as measured by the Patient Global Impression of Change (PGIC) | 3 years
  The Patient Global Impression of Change (PGIC) is used to assess any change in their fibromyalgia since beginning the clinical trial. The PGIC asks patients to describe the change in activity limitations, symptoms, emotions, and overall quality of life on a scale from 0 to 7 since the start of the trial. A score of 0 is characterized by "no change (or condition has gotten worse)" and 7 is characterized by "a great deal better, and considerable improvement that has made the difference", thus, a higher score indicates overall improvement. The PGIC also asks patients to score the degree of change since beginning care at the clinic from 0 to 10. A score of 5 represents no change, while 0 represents "much better" and 10 represents "much worse", thus, a lower score on this question demonstrates a better outcome. These two scores are reviewed separately.
Intensity of specific symptoms pertaining to fibromyalgia, as measured by the Revised Fibromyalgia Impact Questionnaire (FIQ-R) | 3 years
  The Revised Fibromyalgia Impact Questionnaire (FIQ-R) measures how fibromyalgia affects quality of life. The FIQ-R asks patients to rate how difficult it is to perform a list of 9 common activities over the previous 7 days on an 11 point scale (ranging from "no difficulty" to "very difficult". The FIQ-R then asks patients to indicate how often their fibromyalgia impacts their quality of life over the last 7 days on an 11 point scale (ranging from "never" to "always"). Finally, the FIQ-R asks patients to assess the severity of their symptoms on an 11 point scale (ranging from no symptoms to extreme symptoms). These three sub-scales are summed to represent an overall FIQ-R score. A lower value for the FIQ-R represents a better outcome (less severe fibromyalgia).

SECONDARY OUTCOMES:
Intensity of Pain, as measured by the Short-Form McGill Pain Questionnaire (SF-MPQ) | 3 years
  The Short-Form McGill Pain Questionnaire (SF-MPQ) is used to assess fibromyalgia symptoms regarding pain. Patients are asked to rate 15 pain related sensations (throbbing, aching, stabbing, etc.) on a scale of 0 ("none") to 3 ("severe"). Patients are then asked to rate overall pain from 0 ("no pain") to 5 ("excruciating"). These scores are summed to give an overall value for pain, where a low score represents a better outcome (low pain).
Severity of symptoms regarding anxiety and depression, as measured by the Hospital Anxiety and Depression Scale (HADS) | 3 years
  The Hospital Anxiety and Depression Scale (HADS) measures symptoms of anxiety and depression in fibromyalgia. Patients are instructed to rank how much they experience a list of 8 symptoms of anxiety and 8 symptoms of depression on a scale of 0 to 3. 0 represents less extreme symptoms and 3 represents very severe symptoms. These 16 questions are summed such that a low score represents a better outcome (less extreme symptoms of anxiety and depression).
Difficulty with cognitive tasks, as measured by the Cognitive Function (CF) scale | 3 years
  The Cognitive Function (CF) scale measures how often patients struggle with a variety of cognitive tasks. The CF scale lists 25 cognitive tasks and asks patients to assess how often they struggle on a 5 point scale from "very often" to "never". These scores are summed, and a total high score represents better cognitive function and thus a better outcome.
Intensity of fatigue, as measured by the Multidimensional Assessment of Fatigue (MAF) Scale | 3 years
  The Multidimensional Assessment of Fatigue (MAF) Scale asks patients 3 questions regarding how intensely they experience fatigue on a scale of 1 (little fatigue) to 10 (severe fatigue). These scores are summed, and a lower total score represents a better outcome.
Severity and frequency of headaches, as measured by the Headache Questionnaire (HQ) | 3 years
  The Headache Questionnaire (HQ) asks a list of 10 questions regarding the severity and frequency of headaches. These scores are summed, and lower score indicates a better outcome (less frequent and severe headaches).
Difficulty regarding sleep, as measured by the Questionnaire Regarding Sleep (QRS) | 3 years
  The Questionnaire Regarding Sleep (QRS) assesses the quality and quantity of sleep each night. Patients are asked 11 questions relating to how much they sleep (recorded in number of hours) and how often they experience poor sleep quality (on a scale of 0 to 4, where 0 represents not at all and 4 represents very often). These scores are reviewed separately. A high score for how much they sleep demonstrates a better outcome (more sleep) and a low score for how often they experience poor sleep quality demonstrates a better outcome (better sleep quality).

CONTACTS AND LOCATIONS:
Locations (1):
- Immunobiology Labs CNY 149, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Faustman Lab Research Website — http://faustmanlab.org/